CLINICAL TRIAL: NCT02261597
Title: Challenging the Inflammatory Response System: Are Individuals With Insomnia More Reactive?
Brief Title: Challenging the Inflammatory Response System in Insomnia Disorder
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Monika Haack, Assistant Professor of Neurology HMS, Beth Israel Deaconess Medical Center
Other Study IDs: 2014P000297
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Insomnia
Keywords: insomnia, inflammation, stress
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Insomnia Disorder: Testing reactivity of stress-related systems to repeated exposure to the cold pressor test (hand immersion into ice-cold water) among participants with a clinical diagnosis of insomnia disorder.
  Interventions: Behavioral: Cold Pressor Test
- Healthy Control: Testing reactivity of stress-related systems to repeated exposure to the cold pressor test (hand immersion into ice-cold water) among healthy participants without a diagnosis of insomnia disorder.
  Interventions: Behavioral: Cold Pressor Test

INTERVENTIONS:
Behavioral: Cold Pressor Test — Repeated immersion of hand in ice-cold water

SUMMARY:
The main purpose of this study is to understand how insomnia (compared to good sleep) may affect the response of the body to a repeated physiological challenge, such as inserting the hand in ice-cold water for several times in a row. In particular, the investigators are interested in the response of markers that can be associated with stress, such as blood pressure and stress hormones.

DETAILED DESCRIPTION:
Sleep is critical for the regulation and maintenance of biological systems, and sleep deficiency, such as insomnia, has been shown to be associated with elevated risks for cardiovascular, metabolic, and mood disorders.

Despite the high prevalence of insomnia in the population, the investigators understanding of the biological consequences of the disorder with respect to inflammatory, autonomic, and stress system markers is limited, and often not consistent.

In addition, insomnia may not only alter the basal activity of these systems, but may change their reactivity to other stressors and challenges. In support of this assumption are findings showing that poor sleep quality in healthy individuals is associated with a stronger biological response to a stressful challenge, such as the cold pressor test. This test involves the immersion of the hand in ice-cold water. It is one of the most commonly used laboratory physiological challenge tests, provoking not only unpleasantness, but also increases in stress and inflammatory markers.

Investigations of such system's reactivity to challenge may elucidate systems abnormalities that the investigators do not capture by only assessing basal system's levels. For example, in patients with rheumatoid arthritis, basal inflammatory levels are normal, but the response to a physiological stress challenge (cold pressor test) is amplified.

To the investigators knowledge, no studies have measured how insomnia may affect the reactivity of biological systems to a stressful challenge, which may serve as an important indicator of system's dysregulation and associated disease risk.

In this light, the primary goal of this proposal will investigate whether stress-related systems are more reactive to a physiological stressful challenge in insomnia disorder compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between the ages 18-55 years
* Blood chemistry in the normal range
* BMI less than or equal to 35

Specific to insomnia group:

* Diagnosis of insomnia disorder based on DSM-V criteria

Specific for control group:

* Good quality and quantity sleep

Exclusion Criteria:

* Active infection/disease.
* History of neurological, chronic pain, immune, cardiovascular, liver/kidney, or metabolic disorder
* History of psychiatric disorders within the last 6 months prior to study start
* Sleep disorders other than insomnia
* Reynaud's disease
* Psychotropic, sleep, or any other medications or herbs interfering with the inflammatory, autonomic, or HPA system in the last 2 weeks prior to study start, except oral contraceptives
* In psychotherapy or any other behavioral interventions at study start
* Donation of blood or platelets within 3 months of hospital visits
* Pregnant/nursing.
* Substance abuse.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Individuals suffering from insomnia disorder
  * Healthy control sleepers
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haack Monika, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Healthy participants without a diagnosis of insomnia disorder visited the CRC for a one-day stay immediately following an overnight sleep screen
- Insomnia Disorder: Participants with the diagnosis of insomnia disorder (according to DSM-V) visited the CRC for a one-day stay immediately following an overnight sleep screen
Period: Overall Study
Arm/Group | Healthy Controls | Insomnia Disorder
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Insomnia Disorder | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Average age and age range for all participants in the study, and for each arm in the study
  years | 26.09 [18 to 47] | 30.27 [18 to 49] | 28.18 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 16 | 12 | 28
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 11 | 16 | 27
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Response to Physiological Challenge- Change in Plasma Levels of IL-6
Description: Inflammatory marker: Change in plasma levels of IL-6 (pg/mL).
Time Frame: Baseline blood was obtained between 11am-12pm and prior to any Cold Pressor Tests (CPTs). Three CPTs were performed, with 1.5 hours between each one. The first CPT was done at 1pm. Blood draws were obtained 20min and 50 min after each CPT.
Population: Data of 3 participants were excluded from analysis due to development of headache or Iv problems in the course of the experimental study day.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Healthy Controls | Insomnia Disorder
Number analyzed (Participants) | 21 | 20
pg/mL
  Baseline | 1.5013 (0.16892) | 2.1626 (0.67566)
  20min after CPT 1: number analyzed (Participants) | 20 | 19
  20min after CPT 1 | 2.5911 (0.49528) | 2.7269 (0.5303)
  50 min after CPT 1: number analyzed (Participants) | 20 | 19
  50 min after CPT 1 | 3.0318 (0.55967) | 2.7556 (0.31272)
  20 min after CPT 2: number analyzed (Participants) | 20 | 19
  20 min after CPT 2 | 3.7131 (0.65019) | 3.8603 (0.53619)
  50 min after CPT 2: number analyzed (Participants) | 20 | 19
  50 min after CPT 2 | 4.2044 (0.64394) | 3.3381 (0.4539)
  20 min after CPT 3: number analyzed (Participants) | 20 | 17
  20 min after CPT 3 | 5.514 (0.82173) | 5.1606 (0.95047)
  50 min after CPT 3: number analyzed (Participants) | 20 | 18
  50 min after CPT 3 | 5.9841 (1.15086) | 4.3278 (0.75218)

2. Primary Outcome: Stress Reactivity to Physiological Challenge- Change in Serum Levels of Cortisol
Description: HPA marker: Change in serum cortisol levels (ug/dL)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/dL
Arm/Group | Healthy Controls | Insomnia Disorder
Number analyzed (Participants) | 21 | 20
ug/dL
  Baseline | 8.9948 (1.00453) | 9.8250 (0.92339)
  20min after CPT 1: number analyzed (Participants) | 20 | 19
  20min after CPT 1 | 10.6695 (0.61099) | 13.95 (1.22551)
  50 min after CPT 1: number analyzed (Participants) | 20 | 19
  50 min after CPT 1 | 8.3255 (0.47898) | 11.0416 (0.95435)
  20 min after CPT 2: number analyzed (Participants) | 20 | 19
  20 min after CPT 2 | 8.448 (0.57976) | 10.9342 (1.13843)
  50 min after CPT 2: number analyzed (Participants) | 20 | 19
  50 min after CPT 2 | 6.452 (0.39262) | 8.6063 (0.98503)
  20 min after CPT 3: number analyzed (Participants) | 20 | 19
  20 min after CPT 3 | 8.7545 (0.71965) | 9.9168 (1.27366)
  50 min after CPT 3: number analyzed (Participants) | 20 | 19
  50 min after CPT 3 | 6.651 (0.40265) | 8.4684 (1.01139)

3. Secondary Outcome: Glucocorticoid Sensitivity- Percentage of IL-6 Positive Monocytes
Description: Percentage of IL-6 positive monocytes following stimulation with LPS (100pg/mL) and varying concentrations of Dexamethasone
Time Frame: Monocytes are only obtained from the baseline blood draw, which occurs at 11am.
Population: Data of 2 participants were excluded from analysis due to development of headache or Iv problems in the course of the experimental study day.
Measure: Mean (Standard Error); unit: Percentage of IL-6 positive monocytes
Arm/Group | Healthy Controls | Insomnia Disorder
Number analyzed (Participants) | 22 | 20
Percentage of IL-6 positive monocytes | 20.659 (2.9058) | 17.250 (1.9317)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 9-hour period for each particpant.
Groups:
- Insomnia Disorder: Participants with the diagnosis of insomnia disorder (DSM-V) visited the CRC for a one-day stay immediately following an overnight sleep screen.
Arm/Group | Healthy Controls | Insomnia Disorder
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT02261597/Prot_SAP_000.pdf